CLINICAL TRIAL: NCT04597112
Title: Effect of Myofascial Release Technique in Patients with Unilateral Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, fatih bali, Lecturer, Istanbul Kent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.1062
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Cervical Radiculopathy; Cervical Radicular Pain; Cervical; Hernia; Cervical Disc Disease; Cervical Disc Herniation; Pain
Keywords: Cervical Radiculopathy; Pain; Radiculopathy; Cervical; Hernia; Myofascial Release; Exercise
MeSH Terms: conditions — Radiculopathy; Hernia; Pain; Motor Activity | interventions — Myofascial Release Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myofascial Release Group (Experimental): Intervention group, who received conventional therapy and myofascial release therapy.All participants will be given conventional treatment 3 days a week for 4 weeks. Conventional treatment will include 20 minutes hotpack, 5 minutes ultrasound, 20 minutes Transcutaneous Electrical Stimulation. In the intervention group, the myofascial release technique will be applied to the wrist flexors and extensors, elbow flexors and extensors, pectoralis, supraspinatus, infraspinatus, trapezius muscles, starting from the fingers after the conventional treatment, 3 days a week for 4 weeks.
  Interventions: Other: Myofascial Release Technique
- Exercise Group (Active Comparator): The control group will consist of patients who received conventional therapy and exercise therapy. All participants will be given conventional treatment 3 days a week for 4 weeks. Conventional treatment will include 20 minutes hotpack, 5 minutes ultrasound, 20 minutes Transcutaneous Electrical Stimulation. After conventional treatment, a program consisting of neck extension, lateral flexion and rotation range of motion, stretching of the trapezius muscles and strengthening of the neck extensor muscles will be applied to the control group in the presence of a physiotherapist 3 days a week for 4 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Myofascial Release Technique — Myofascial release focuses on reducing pain by easing the tension and tightness in the trigger points. Therapist will gently massage the myofascia and feel for stiff or tightened areas. Normal myofascia should feel pliable and elastic. The therapist will begin massaging and stretching the areas that feel rigid with light manual pressure. The therapist then aids the tissue and supportive sheath in releasing pressure and tightness. The process is repeated multiple times on the same trigger point and on other trigger points until the therapist feels the tension is fully released.
  Arms: Myofascial Release Group
Other: Exercise — Exercise is recommended by physical therapists for most cervical radiculopathy patients.
  In this study, a customized exercise program will be applied for patients with cervical radiculopathy.
  Arms: Exercise Group

SUMMARY:
The aim of the study is to investigate the effectiveness of myofascial release technique on pain, range of motion, muscle strength, functionality and quality of life in individuals diagnosed with cervical radiculopathy with unilateral arm involvement and compare this with exercise. The individuals included in the study will be randomized into two groups, 17 control and 17 study groups. Sessions will be 3 days a week for 4 weeks. Conventional physiotherapy and exercise program will be applied to the control group, conventional physiotherapy and myofascial release technique will be applied in the intervention group. Conventional physiotherapy methods; It will include Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound (US), hotpack agents. Exercise program; extension, right and left lateral flexion, right and left rotation exercises, chin-tuck, right and left upper trapezius muscle group stretching, neck extensor muscle group isometric strengthening exercises. Myofascial release will be applied to the fingers, wrist flexor-extensor muscle groups, elbow flexor-extensor muscle groups, pectoral muscles and rotator cuff muscle groups. Patients will be evaluated before and after treatment with Visual Analogue Scale (VAS), Goniometric measurements, algometer, myometer, Neck Disability Scale, "Disability of Arm, Shoulder and Hand" Questionnaire (DASH).

ELIGIBILITY:
Inclusion Criteria:

* Getting a diagnosis of cervical radiculopathy
* Unilateral upper extremity symptoms at least for a month
* The diagnosis is confirmed by the medical board report
* Being between the ages of 30-65
* Voluntary acceptance to participate in the study

Exclusion Criteria:

* Previous cervical surgery
* Previous cervical trauma
* Have had myofascial therapy or conventional therapy for cervical radiculopathy
* Long-term use of corticosteroids
* Congenital torticollis history
* Using nonsteroidal anti-inflammatory drugs for long time
* Migraine
* Cancer
* Tumor
* Osteoporosis
* Pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Algometer | 10 minutes
  It is a device used to evaluate the sensitivity to pain and to determine the perception of pressure. The pressure algometer has proven useful in evaluating fibrositis and hypersensitive spots, trigger points, arthritis activation, and visceral pain-pressure sensitivity.
Myometer | 10 minutes
  Hand myometer is a means of expressing force quantitatively. It is preferred over other dynamometers because of its ease of use and portability.
Electrogoniometer | 10 minutes
  It is an evaluation tool used to record the objective measurement of joint range of motion.
Visual Analog Scale | 1 minutes
  Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically into digital. Two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line and the patient is asked to indicate where his / her condition is appropriate by drawing a line or by placing a dot or marking.

SECONDARY OUTCOMES:
Neck Disability Index | 10 minutes
  It is a test consisting of ten parts that determines to what extent neck pain affects daily life activities. The questions are of a nature that includes the intensity of pain and the effect of pain on occupational and social activity and its relationship with emotional factors. 10 cm visual analogue scale (VAS) is used for each question. High scores indicate the severity of the disease.
Disability of Arm Shoulder and Hand Test | 10 minutes
  This questionnaire evaluates the disability and activity limitations resulting from upper extremity injury, as well as the restriction of leisure activities and work participation. The DASH questionnaire consists of three parts. According to the survey results; A result of 0-100 is obtained from each section. (0 = no apology, 100 = maximum apology).

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Bali, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No